CLINICAL TRIAL: NCT03854318
Title: Longitudinal Studies of Patients and Families With Familial Platelet Disorders With Associated Myeloid Malignancy (FPDMM) Caused by RUNX1 Germline Variants or FPDMM-Like Conditions
Brief Title: Longitudinal Studies of Patient With FPDMM
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190059; 19-HG-0059
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-21

CONDITIONS: Inherited Hematological Diseases; Rare Diseases; FPDMM
Keywords: inherited hematological diseases; Rare Diseases; Hematological Malignancies; Cancer; Acute Myeloid Leukemia; Natural History
MeSH Terms: conditions — Rare Diseases; Platelet Disorder, Familial, with Associated Myeloid Malignancy; Hematologic Neoplasms; Neoplasms; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Family: Direct family members of enrolled patients will be asked to enroll in the study to provide specimens for genetic testing, next-generation sequencing, and other related studies.
- RUNX1: Patients enrolled in this protocol will have been referred with a known or suspected RUNX1 mutation.

SUMMARY:
Background:

Genes tell the body and its cells how to work. Familial platelet disease (FPD) or FPD with associated malignancies (FPDMM) is caused by a variant in the gene RUNX1. People with this disease may have problems with their blood and bleed for a long time when they are injured. Researchers want to learn more about RUNX1 variants and FPD.

Objective:

To learn more about FPD in people with RUNX1 variants to lead to better diagnosis, monitoring, and treatment.

Eligibility:

People any age with a suspected or confirmed RUNX1 variant

People who have a family member with the variant

Design:

All participants will be screened with a phone call and a blood, saliva, or cheek cell sample.

Participants with a suspected or confirmed variant will have 1 visit. It will last about 2 days. They will then have visits at least once a year.

Visits will include:

* Medical history and physical exam
* Blood tests or saliva sample
* Possible skin biopsy: A small piece of the participant s skin will be removed.
* Bone marrow aspiration or biopsy: The participant s bone marrow will be removed by needle from a large bone such as the hip bone.
* Possible apheresis: Blood will be removed from the body and certain blood cells will be taken out. The rest of the blood is returned to the body.

Between visits, participants with a suspected or confirmed variant will keep a diary of disease symptoms and signs.

Samples from all participants may be used for genetic testing

DETAILED DESCRIPTION:
Study Description:

This is a natural history study of patients with familial platelet disorder with associated myeloid malignancies (FPDMM), also known as FPD and FPDAML, who undergo diagnostic clinical tests, diagnostic genetic tests, and yearly follow-up visits; and the collected biological samples will be used for biomedical research to understand the disease mechanism, including genomic sequencing. Unaffected family members will participate and serve as controls for studies of the affected family members.

Objectives:

Primary Objective: To identify and follow patients with germline variants in the RUNX1 gene, which leads to FPDMM, an autosomal dominant disorder, with the hope of identifying biomarkers that can predict which patients will progress and develop malignancies, as well as the timing of the progression and the severity of the malignancies.

Secondary Objectives: To identify secondary gene mutations that may impact clinical presentation, disease severity, and progression to malignancies. Secondary gene discovery will distinguish subpopulations of patients and may inform clinical care and improve diagnosis. To profile non-hematopoietic presentations of FPDMM. To identify genetic basis for patients with FPDMM-like clinical presentation but without known RUNX1 variants. To longitudinally assess psychosocial experiences, psychosocial functioning, and health related quality of life of persons living with RUNX1-FPD.

Exploratory Objective: Identify new therapeutic strategies.

Endpoints:

Primary Endpoint: The primary endpoint is progression to malignancy in patients with FPD (FPDMM). Patients who develop malignancies will continue in the study for longitudinal observation.

ELIGIBILITY:
* INCLUSION CRITIERIA:

Patients enrolled in this protocol will have been referred with a known or suspected variant in the RUNX1 gene. Patients with suspected RUNX1 variants are those with clinical features of FPD but who have not been tested for RUNX1, or who were negative on standard testing. The Principal Investigator, along with consulting specialists, will review the medical records of prospective patients and offer enrollment based upon the potential to help the individual, to learn from the patient, or to initiate clinical or basic research suggested by the patient's workup. Persons interested in participation may be given a screening questionnaire to determine eligibility. The questions about hematologic manifestations in the screening questionnaire are important to help us determine if RUNX1 variants are likely to be pathogenic, or if there is a high clinical suspicion of RUNX1 (abnormal platelets, bleeding, bruising, leukemia etc.). Unaffected family members may be asked to enroll in the study to provide specimens (saliva, blood, skin) for genetic testing, next-generation sequencing, and other related studies. Enrolled subjects can be any sex and any age. There are no upper or lower age restrictions on this study.

EXCLUSION CRITIERIA:

There are no exclusionary criteria.

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients (and direct family members of patients) enrolled in this protocol will have been referred with a known or suspected RUNX1 mutation.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Natural History | Ongoing
  This protocol continues the decades-long tradition of identifying and examining patients with rare genetic diseases and characterizing the natural history.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Liu, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
pending
Supporting Information: Study Protocol
Time Frame: pending
Access Criteria: pending

REFERENCES:
- [Derived] Kajdic A, Deuitch NT, Bresciani E, Chong SN, Craft KM, Davis J, Bashtawi R, McReynolds LJ, Giri N, Young DJ, Liu PP. Hematologic malignancies in pediatric patients with RUNX1-Familial Platelet Disorder with Associated Myeloid Malignancy. Blood Adv. 2026 Jan 30:bloodadvances.2025017808. doi: 10.1182/bloodadvances.2025017808. Online ahead of print. PMID 41616279
- [Derived] Yu K, Deuitch N, Merguerian M, Cunningham L, Davis J, Bresciani E, Diemer J, Andrews E, Young A, Donovan F, Sood R, Craft K, Chong S, Chandrasekharappa S, Mullikin J, Liu PP. Genomic landscape of patients with germline RUNX1 variants and familial platelet disorder with myeloid malignancy. Blood Adv. 2024 Jan 23;8(2):497-511. doi: 10.1182/bloodadvances.2023011165. PMID 38019014
- [Derived] Cunningham L, Merguerian M, Calvo KR, Davis J, Deuitch NT, Dulau-Florea A, Patel N, Yu K, Sacco K, Bhattacharya S, Passi M, Ozkaya N, De Leon S, Chong S, Craft K, Diemer J, Bresciani E, O'Brien K, Andrews EJ, Park N, Hathaway L, Cowen EW, Heller T, Ryan K, Barochia A, Nghiem K, Niemela J, Rosenzweig S, Young DJ, Frischmeyer-Guerrerio PA, Braylan R, Liu PP. Natural history study of patients with familial platelet disorder with associated myeloid malignancy. Blood. 2023 Dec 21;142(25):2146-2158. doi: 10.1182/blood.2023019746. PMID 37738626
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-HG-0059.html